CLINICAL TRIAL: NCT00407472
Title: ATS-1 Needle Free Injection Device Study-a Device for Administering r-hGH (Saizen) to Treat Growth Hormone Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 25821
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: Bio-equivalence study in healthy volunteers, indication; of product is growth hormone deficiency

INTERVENTIONS:
Device: ATS-1 needle free device

SUMMARY:
This study was a Phase I, open label, randomized, 2-period, 2-sequence, crossover study designed to assess the relative bioavailability of Saizen administered by the ATS-1 needle-free injection device and a standard needle and syringe. Informed consent was obtained prior to screening. All screening assessments establishing subject eligibility were performed in the 21 days before dosing. Randomization Pre-dose on Day 1, subjects were randomized to one of the two treatment sequences: Sequence 1: SC Saizen administered by the Standard needle and syringe (Period 1) followed by the administration using the ATS-1 device (Period 2). Sequence 2: SC Saizen administered by the ATS-1 device (Period 1) followed by administration using the standard needle and syringe (Period 2).

Subjects were resident at the Unit from approximately 19:00 on Day -1 until Day 2 (approximately 30 hours (h) post dose) of each treatment period. An IV Stilamin infusion was commenced 1 h before. Saizen administration and stopped immediately after the last pharmacokinetic (PK) blood sample has been taken, i.e. a 25 h infusion. Stilamin was administered as a constant IV infusion at a rate of approximately 118 mg/h (40 mL/h), which corresponds to 1.65 mg/kg body weight/h for a person weighing 70kg. Dosing with Saizen occurred between approximately 0800 and 0900 h on Day 1 of each treatment period after an overnight fast of at least 10h. Subjects were dosed with Saizen at the same time on Day 1 in Periods 1 and 2. There was a minimum of 7-day washout between treatment periods 1 and 2.

Laboratory safety tests, ECGs were taken at protocol specified time points and blood samples for the assessment of glucose and growth hormone were taken immediately predose and 1, 2, 3, 4 4.5, 5, 5.5, 6, 7, 8, 12, 18 and 24 h post dose. A post-study visit took place 33+/- 3 days after dosing a treatment period 2.

ELIGIBILITY:
Inclusion Criteria:

* Male Subjects age 21 to 50
* Have given written informed consent
* Have a body weight greater than 60 kg and a body mass index (BMI) in the range of 22 30 (BMI - weight (kg) / height (m) 2)
* Have vital signs in the following normal range:
* Oral body temperature: 35.0 - 37.5 0C
* Blood Pressure (BP): Supine BP after at least 3 minutes of supine rest Systolic BP: 90 - 150 mm Hg, diastolic P: 50 - 95 mm Hg, Supine heart rate after at least 3 minutes of rest: 40 - 90 bpm
* Be non-smoker or smoke less than or equal to five cigarettes (or use an equivalent amount of tobacco per day and be willing not to smoke whilst resident in the clinical unit
* Be able to communicate well with the Principal Investigator and be willing to comply with the requirements of the entire study
* Agree to use barrier contraception (condom and spermicide) during the study and for three months following completion of the post study visit.

Exclusion Criteria:

* Existence of any surgical or medical condition which in the opinion of the Principal Investigator might interfere with the absorption, distribution, metabolism or elimination of the investigational medicinal product or with the aims of the study
* Have any clinically significant abnormality in the results of the screening safety laboratory tests
* Have an clinically significant abnormality on the 12-lead resting ECG at screening
* Have positive results from virology examination for Hepatitis surface antigen (HBsAg) (not due to vaccination), Hepatitis C Virus (HCV) and Human Immunodeficiency Virus (HIV 1 and 2) at screening
* History or presence of hypertension or other significant cardiovascular abnormalities
* History or presence of cholelithiasis
* Significant history or clinical evidence of auto-immune, gastrointestinal, hematological, haemaoppoietic, hepatic, neurological, pancreatic or renal disease
* History or presence of diabetes
* Definite or suspected personal history or family history of adverse drug reaction or hypersensitivity to drugs with similar chemical structure to somatotropin or somtostatin
* Use of any chronic medication
* Presence or history of any serious allergy (requiring hospitalization or prolonged systemic treatment)
* History or presence of drug or alcohol abuse. The limits of alcohol consumption for inclusion in the study are defined as an average daily intake of 3 units or a maximum weekly intake of grater than 21 units (1 unit equals 340 mL of beer, 115 mL of wine or 43 mL or spirits)
* Loss or donation or more than 400 mL of blood in the 12 weeks before dosing
* Subjects who have used any prescription drugs within 2 weeks or over-the-counter medication (with the exception of paracetamol and multi-vitamins) within 1 week before dosing without prior approval from the investigator
* Administration of any investigational drug in the 12 weeks before dosing

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38
Dates: Start 2005-09; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Priestley, MBChB MFPM, Principal Investigator — Bourn Hall Clinic

REFERENCES:
- See also: Full FDA approved prescribing information can be found here — http://www.saizenus.com